CLINICAL TRIAL: NCT05106322
Title: Estimation of Steatosis on Liver Transplants by Intraoperative Spectrometry
Acronym: iGRAISSE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210949
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Liver Transplants
Keywords: macrosteatosis; spectrometry; liver transplantation; biopsy; primary non-function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplants: Whole liver transplants proposed for organ harvesting from brain-dead donors and assigned by the Biomedicine Agency.
  Interventions: Other: intraoperative spectrometer scan

INTERVENTIONS:
Other: intraoperative spectrometer scan — intraoperative spectrometer scan (five scans on the left lobe) before clamping the aorta

SUMMARY:
The goal is to have a small spectrometer (pocket size) , reliable and rapid tool that can be used during liver harvesting, which enables macrosteatosis to be evaluated reproducibly and selectively, at any time.

This tool must be minimally invasive, inexpensive and without significantly impacting the general organization of multi-organ harvesting.

In the operating room, the surgeon will perform an intraoperative spectrometer scan (five scans on the left lobe) before clamping the aorta. The surgeon will not be informed of the results of the spectrometer, and will carry out (or not) the biopsy. The spectrometers' results will be compared with definitive histological findings.

ELIGIBILITY:
Inclusion Criteria:

* Brain-dead donor
* Age ≥18 years old
* No restriction on the part of the donor or his family regarding the use of the data for research purposes.
* No fibrous appearance of the graft (visual assessment), corresponding to a Metavir score ≥ F2

Exclusion Criteria:

* Living donor
* Donor within the Maastricht III criteria (cardiac arrest)
* Pre-existing hepatic injury / trauma preventing the intraoperative use of the pocket spectrometer
* History of supra-mesocolic surgery or peritonitis leading to perihepatic adhesions (preventing the use of pocket spectrometer)
* History of chemotherapy -- Biological cholestasis:

  * GGT> 400 IU / L
  * or total bilirubin ≥ 60micromol / L
  * or conjugated bilirubin ≥ 30micromol / L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Whole liver transplants proposed for organ harvesting from brain-dead donors assigned by the Biomedicine Agency
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Evaluate the concordance between the macrosteatosis quantified by the pocket spectrometer and the macrosteatosis content evaluated by the standard pathological analysis | J0 = intraoperative
  Agreement (intra-class correlation coefficient) between the% of macrosteatosis estimated by the pocket spectrometer and that quantified by the pathologist on biopsy (final results only)

SECONDARY OUTCOMES:
Evaluation of the spectrometer performance for diagnosis to detect macrosteatosis> 30% and> 60% taking the pathology as a reference standard | J0 = intraoperative
  Area under the ROC curve (AUC), sensitivity, specificity, likelihood ratio and predictive values of the spectrometer to detect macrosteatosis> 30% and> 60%
Assessment of the technical feasibility of using the spectrometer in daily practice, analysis of the causes and incidence of failures (technical or organizational) | J0 = intraoperative
  Number of time where the measurement by the pocket spectrometer was successful, ie where it was possible to perform the scans and obtain an estimate of the macrosteatosis, and description of the causes for failure.
Estimation of the concordance between the macrosteatosis values provided by the frozen section analysis, if performed, and the definitive pathology and comparison with the concordance of the pocket spectrometer estimated for the primary objective | J0 = intraoperative
  Agreement (intra-class correlation coefficient) between the% of macrosteatosis estimated by the pathologist extemporaneously when performed and te one quantified by the pathologist on biopsy (final results only).
Assessment of the concordance between the macrosteatosis visually assessed by the harvesting surgeon and the definitive pathological data | J0 = intraoperative
  Agreement (kappa coefficient) between the% of macrosteatosis macroscopically estimated by the pathologist (in 3 categories: 0-30%, 31-60%,> 60%) and that quantified by the pathologist on biopsy (final results only )
Evaluation of the potential impact of spectrometer results on the surgeon's decision to accept the graft using simulated results | J0 = intraoperative
  Percentage of acquisitions where the operator would have modified his decision (accept / reject the graft) if the spectrometer estimate had been communicated (scenarios simulated in the questionnaires)
Modification and improvement of the current algorithm based on the spectra of the entire cohort in order to assess the gain in "spectrometer - anatomopathology" | J0 = intraoperative
  Agreement (intra-class correlation coefficient) between the percentage of macrosteatosis estimated by the spectrometer using the second version of the algorithm and the macrosteatosis quantified by pathology
Attempt to create a microsteatosis prediction algorithm (version 3) using data from the global cohort | J0 = intraoperative
  Agreement (intra-class correlation coefficient) between the percentage of microsteatosis estimated by the spectrometer and the microsteatosis quantified by the pathology

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GOLSE, Principal Investigator — APHP
Locations (3):
- France (3):
  - Centre Hépato Biliaire de l'hopital Paul Brousse, Villejuif
  - Hôpital Beaujon, Clichy, Île-de-France Region
  - Hôpital Pitié-Salpetriere, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No